CLINICAL TRIAL: NCT06369792
Title: EVALUATION PROSPECTIVE DE L'AIDE AU DIAGNOSTIC ET AU TRAITEMENT PAR BIOMARQUEURS SANGUINS CHEZ DES PATIENTS DRUG-NAÏFS AMBULATOIRES SOUFFRANT DE DEPRESSION
Brief Title: PROSPECTIVE EVALUATION OF BLOOD BIOMARKERS AS AN AID TO DIAGNOSTIC AND TREATMENT IN DRUG-NAIVE PATIENTS WITH DEPRESSION
Status: Recruiting | Type: Observational
Sponsor: Les Toises - Psychiatry and Psychotherapy Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00266
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder; Bipolar Disorder; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational (non-interventional) prospective study, carried out in drug-naïve outpatients who start a treatment with escitalopram, fluoxetine, sertraline or quetiapine. Five blood samples are collected (i.e. before initiating the drug, and then after 1, 2, 4 and 8 weeks of treatment). It does not affect the choice or the treatment dose. The primary objective of this study is to measure the association between the EDIT-B® editing signature and response to pharmacological treatment in drug-naïve patients. Results of this research could provide an aid to early diagnosis, optimize pharmacological treatment and guide clinical practice towards individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult drug-naïve outpatients suffering from depression and/or bipolar disorders who start a pharmacological treatment with escitalopram, fluoxetine, sertraline or quetiapine and who gave his written informed consent to participate in the present study.

Exclusion Criteria:

* Any patient without capacity of discernment or with harmful use of psychoactive substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes drug-naïve adult outpatients (aged 18 or over) with depression (F32-33) and/or bipolar disorder (F30-F31) who start escitalopram, fluoxetine, sertraline or quetiapine.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
psychiatric symptomatology | At baseline, 1,2,4,8 weeks
  self- and hetero-questionnaire psychiatric scales
EDIT-B profiling | At baseline, 1,2,4,8 weeks
  Measurement of RNA editing over time

CONTACTS AND LOCATIONS:
Locations (1):
- Les Toises - Psychiatry and Psychotherapy Center, Lausanne, Switzerland